CLINICAL TRIAL: NCT01682070
Title: A Randomized, Double-blind, Placebo-controlled Study to Determine Safety, Tolerability and the Optimal Effective Dose of SUBLIVAC FIX Phleum Pratense in Patients With Allergic Rhinitis/Rhinoconjunctivitis Caused by Grass Pollen
Brief Title: SUBLIVAC FIX Phleum Pratense DT/DRF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP/0036
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Allergic Rhinitis; Allergic Rhinoconjunctivitis
Keywords: Sublingual immunotherapy; Dose range finding; Dose tolerability; grass pollen; Allergic rhinitis/rhinoconjunctivitis; Safety; Immunogenicity
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- SUBLIVAC FIX Phleum prat. 0 AUN/ml (Placebo Comparator)
  Interventions: Biological: Placebo
- SUBLIVAC FIX Phleum prat. 3,333 AUN/ml (Experimental)
  Interventions: Biological: SUBLIVAC FIX phleum prat.
- SUBLIVAC FIX phleum prat. 10,000 AUN/ml (Experimental)
  Interventions: Biological: SUBLIVAC FIX phleum prat.
- SUBLIVAC FIX phleum prat. 20,000 AUN/ml (Experimental): Evaluation of the SUBLIVAC FIX Phleum prat. 20,000 AUN/ml by an independent safety committee
  Interventions: Biological: SUBLIVAC FIX phleum prat.
- SUBLIVAC FIX Phleum prat. 40,000 AUN/ml (Experimental): Start of SUBLIVAC FIX Phleum prat. 40,000 AUN/ml arm depends on safety in the SUBLIVAC FIX Phleum prat. 20,000 AUN/ml arm evaluated by an independent safety committee
  Interventions: Biological: SUBLIVAC FIX phleum prat.

INTERVENTIONS:
Biological: SUBLIVAC FIX phleum prat. — Comparison of different dosages to placebo
  Arms: SUBLIVAC FIX Phleum prat. 3,333 AUN/ml; SUBLIVAC FIX Phleum prat. 40,000 AUN/ml; SUBLIVAC FIX phleum prat. 10,000 AUN/ml; SUBLIVAC FIX phleum prat. 20,000 AUN/ml
Biological: Placebo
  Arms: SUBLIVAC FIX Phleum prat. 0 AUN/ml

SUMMARY:
The aim of the study is to determine the optimal effective dose of SUBLIVAC FIX Phleum pratense based on reduction of upper airways reactivity after 5 months of treatment with different dosages of SUBLIVAC FIX Phleum pratense compared to placebo. Furthermore, safety and tolerability will be assessed by the number of related Adverse Events of different dosages of SUBLIVAC FIX Phleum pratense compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 ≤ 60 years
* Allergic rhinitis/rhinoconjunctivitis related to grass pollen with or without concomitant mild to moderate persistent asthma
* FEV1 > 70% for patients with a history of asthma, FEV > 70% or PEF > 80% for patients without a history of asthma
* A positive SPT (mean wheal diameter ≥ 3mm compared to negative control and negative control should be negative) for grass pollen assessed within 1 year before randomization.
* Positive serum specific anti-grass IgE-test (> 0.7 U/mL)
* A positive TNPT for grass pollen at screening (Lebel score ≥ 6) at ≤10,000 AU/mL

Exclusion Criteria:

* Patients with (expected) clinically relevant symptoms during the course of the trial due to concomitant sensitization i.e. positive SPT (mean wheal diameter ≥ 3mm) to allergens other than grass pollen
* Patients sensitized to pets should not be included if they are regularly exposed to pets and are symptomatic upon exposure to pets
* Completed immunotherapy (SCIT or SLIT) with grass pollen allergens within the past 5 years
* Completed unsuccessful specific immunotherapy in the past
* Vaccination within one week before start of therapy or during the initiation phase
* Anti-IgE therapy within the 6 months prior to inclusion and during the study
* Severe immune disorders (including auto-immune diseases) and/or diseases requiring immunosuppressive drugs
* Active malignancies or any malignant disease during the previous 5 years
* Severe uncontrolled diseases that could increase the risk for patients participating in the study, including but not limited to: cardiovascular insufficiency, any severe or unstable lung diseases, endocrine diseases, clinically significant renal or hepatic diseases, or haematological disorders
* Active inflammation or infection of the target organs (nose, eyes or lower airways) at the start of the study
* Moderate to severe nasal obstructive diseases that preclude a TNPT (septal deviation, nasal polyps, recent nasal surgery, etc.)
* Diseases with a contraindication for the use of Adrenaline (e.g. hyperthyroidism, glaucoma)
* Use of systemic steroids within 4 weeks before start of the study and during the study
* Treatment with systemic and local β-blockers
* Participation in a clinical study with a new investigational drug within the last 3 months or for a biological within the last 6 months prior to or during the study
* Pregnancy, lactation or inadequate contraceptive measures for women of child-bearing age (adequate contraceptive measures will be the use of a contraceptive device or -pill)
* Alcohol, drug or medication abuse within the past year
* Any clinically significant abnormal laboratory parameter at screening
* Lack of cooperation or compliance
* Severe psychiatric, psychological, or neurological disorders
* Patients who are employees of the institution or 1st grade relatives or partners of the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 266 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Nasal Provocation Test (NPT) | 5 months
Number of related AEs | First ten days of study medication intake

SECONDARY OUTCOMES:
Serum specific immunoglobulin levels (IgE, IgG, IgG4) | 5 months
Number of local and systemic reactions | Duration of study medication intake (approximately 5 months)
Peak Nasal Inspiratory Flow (PNIF) | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Walter G. Canonica, Prof. Dr., Study Chair — Allergy and Respiratory Diseases University of Genoa
Locations (23):
- Germany (11):
  - CIMS Studienzentrum Bamberg, Bamberg
  - Charité Universitaetsmedizin Berlin Klinik f. Dermatalogie, Venerologie u. Allergologie, Campus Charité Mitte, Berlin
  - Klinik u. Poliklinik f. Dermatologie u. Allergologie Universität Bonn, Bonn
  - Dermatologikum Hamburg - Dept. of Allergology, Hamburg
  - HNO Praxis Dr. Horn/Dr. Zeuner, Heidelberg
  - Klinikum der Johann-Wolfgang-Goethe Universität - Zentrum f. Kinder- u. Jugendmedizin, Hessen
  - Dres.Ina Röhrig-Petering und Holger Petering, Hildesheim
  - FÄ HNO Allergologie, Saalfeld
  - Klinikum Stuttgart - Klinik f. Dermatologie u. Allergologie, Stuttgart
  - Universitäts- Hautklinik Eberhard Karls - Universität Tübingen Department of Dermatology, Tübingen
  - Dr. Med. Ulrich Neumann, Wolmirstedt
- Poland (12):
  - Prywatna Praktyka Lekarska Gabinet Pediatryczno-Alergologiczny, Bialystok
  - SP-ZOZ Ośrodek Zdrowia w Bieńkówce, Bieńkówka
  - NZOS "Zdrowie", Cieszyn
  - Poradnia Alergologiczna Samodzielnego Publicznego Szpitala Nr 5 Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Poradnia Alergologii i Chorób Płuc SP ZOZ Uniwersytecki Szpital Kliniczny im Norberta Barlickiego w Łodzi, Lodz
  - NZOZ Centrum Alergologii, Lodz
  - ALERGOPNEUMA Marek Michnar i Wspolnicy Sp. Jawna, Lublin
  - NZOZ Centrum Alergologii, Lublin
  - Centrum Alergologii Teresa Hofman, Poznan
  - ALERGOMED Specjalistyczna Przychodnia Lekarska Sp. z o.o., Tarnów
  - EMC Intytut Medyczny S.A. Przychodnia przy Łowieckiej, Wroclaw
  - NZOZ Lekarze Specjaliści J. Małolepszy i Partnerzy, Wroclaw